CLINICAL TRIAL: NCT04775433
Title: 'The Actual and Perceived Levels of Physical Fitness and Lifestyle Habits in University of Malta Students'
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Malta (Other)
Responsible Party: Principal Investigator, Mary Grace Grima, Principal Investigator, Physiotherapy Clinician, University of Malta
Other Study IDs: UniMalta
Record Dates: First submitted 2021-02-08; First posted 2021-03-01 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Physical Fitness; Lifestyle, Healthy
Keywords: perceived,; physical fitness; lifestyle habits; alcohol consumption; sleep; tobacco smoking
MeSH Terms: conditions — Alcohol Drinking; Tobacco Smoking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ultimate goal for every health-care system is to have a healthy population by maintaining good physical fitness levels and lifestyle habits, including regular physical activity, good sleep quality, smoking and alcohol abstinence. The main components of physical fitness include body composition, muscular strength and endurance, flexibility and cardiovascular endurance. National research based on actual and perceived physical fitness levels in University of Malta (UM) students where both physical and non-physical testing are included, is lacking.

Also, to the knowledge of the researcher, no such research investigated the relationship between the actual and perceived levels of physical fitness with lifestyle habits (smoking, alcohol consumption and sleep).

This study aims to investigate the correlation between the actual and perceived levels of physical fitness (body composition, cardiovascular endurance, muscular strength and endurance and flexibility) by physical and non-physical testing, the correlation between lifestyle patterns (smoking, alcohol consumption and sleep.

DETAILED DESCRIPTION:
The ultimate goal for every health-care system is to have a healthy population by maintaining good physical fitness levels and lifestyle habits, including regular physical activity, good sleep quality, smoking and alcohol abstinence. The main components of physical fitness include body composition, muscular strength and endurance, flexibility and cardiovascular endurance. A national research based on actual and perceived physical fitness levels in University of Malta (UM) students where both physical and non-physical testing are included, is lacking.

Also, to the knowledge of the researcher, no such research investigated the relationship between the actual and perceived levels of physical fitness with lifestyle habits (smoking, alcohol consumption and sleep).

This study aims to investigate the correlation between the actual and perceived levels of physical fitness (body composition, cardiovascular endurance, muscular strength and endurance and flexibility) by physical and non-physical testing, the correlation between lifestyle patterns (smoking, alcohol consumption and sleep.

This proposed research shall adopt a quantitative-based, correlational type of study design. Registrar and student organisations shall act as intermediary entities and send an information letter via electronic mail to all students aged between 18-30 years. All participants who respond to the call, on attendance to a pre-set date for a face-to-face information session by the researcher, will be asked to sign an informed consent form. Each participant will come for data collection only once at the Department of Physiotherapy laboratories, Faculty of Health Sciences, at the University of Malta and shall take around 20 minutes.

Every query will be answered, a detailed explanation and demonstration of each test will be given to each participant, and qualified physiotherapists will perform the testing.

In this proposed study, the aim of The Fagerstrom Test for Nicotine Dependence (FTND), Alcohol Use Disorders Identification Test (AUDIT) and Pittsburgh Sleep Quality Index (PSQI) is to quantitatively study various lifestyle habits in UM students including smoking, alcohol consumption and sleep quality respectively. The Self-Perceived Fitness questionnaire (SPF) shall be used to measure self-perceived physical fitness in University of Malta students. The Fagerstrom Test for Nicotine Dependence is open-access, and can be used for free for research purposes. On the other hand, permissions to use the Alcohol Use Disorders Identification Test, Pittsburgh Sleep Quality Index and Self-Perceived Fitness questionnaire were given by their respective authors.

Body composition shall be measured by Body Mass Index and Waist Circumference, lower and upper limb flexibility shall be measured by Modified Sit and Reach Test and Back Scratch Test respectively. In addition, cardiovascular endurance shall be measured by Resting Heart Rate, Blood Pressure and 3 Min Step Test, while Squats and Push-ups until fatigue shall be used to measure lower and upper limb muscular strength and endurance. All data will then be analysed using statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* all students aged between 18-30 years, and enrolled within the University of Malta in 2021-2022

Exclusion Criteria:

* Participants who underwent any orthopaedic surgery/trauma in the previous two years or who suffer from hereditary diseases that may lead to movement restrictions, compromised muscular strength, endurance or flexibility, since any of these may limit generalisability of results.
* Participants who are taking medications that cause tachycardia, suffer from resting angina, uncontrolled respiratory conditions, diabetes and high blood pressure.

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: All university of Malta students, both males and females, and aged between 18-30 years, shall be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Alcohol Consumption | through study completion, an average of 1 year.
  Alcohol Use Disorders Identification Test (AUDIT)
Tobacco Smoking | through study completion, an average of 1 year.
  Fagerstrom Test for Nicotine Dependence
Sleeping Pattern and Quality | through study completion, an average of 1 year.
  Pittsburgh Sleep Quality Index
Perceived Physical Fitness | through study completion, an average of 1 year.
  Self-perceived fitness Questionnaire
Physical Fitness- Body Composition | through study completion, an average of 1 year.
  Waist Circumference
Physical Fitness- Body Composition | through study completion, an average of 1 year.
  Body Mass Index
Physical Fitness- Flexibility | through study completion, an average of 1 year.
  Modified Sit and Reach Test
Physical Fitness- Flexibility | through study completion, an average of 1 year.
  Back Scratch Test
Physical Fitness- Muscular strength and endurance | through study completion, an average of 1 year.
  Squats until fatigue
Physical Fitness- Muscular strength and endurance | through study completion, an average of 1 year.
  Push-Ups until fatigue
Physical Fitness- Cardiovascular Endurance | through study completion, an average of 1 year.
  Resting Heart Rate (RHR)
Physical Fitness- Cardiovascular Endurance | through study completion, an average of 1 year.
  Blood Pressure (BP)
Physical Fitness- Cardiovascular Endurance | through study completion, an average of 1 year.
  3 Minute Step Test

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Lab, Physiotherapy Department, Faculty of Health Sciences, Mater Dei Hospital, Msida, Malta

IPD SHARING:
Plan to Share IPD: No